CLINICAL TRIAL: NCT04362618
Title: Exercise Therapy for Osteoarthritis Pain: How Does it Work?
Acronym: KOA-PAIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Collaborators: Universitair Ziekenhuis Brussel (Other); AZ St.-Dimpna Geel (Other)
Responsible Party: Principal Investigator, Prof. Ivan Bautmans, Prof. dr., Vrije Universiteit Brussel
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: G040919N_KOA_PAIN
Record Dates: First submitted 2020-02-28; First posted 2020-04-27 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Knee Osteoarthritis
Keywords: Osteoarthritis; Exercise; Acute effects; Inflammation; Endogenous hypoalgesia
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Motor Activity; Inflammation

STUDY DESIGN:
Intervention Model Description: The patients will be randomly allocated to 12 weeks of either muscle strengthening training (MST), behavioural graded activity (BGA) or control. Randomization will be performed by using the method of randomly permuted blocks, utilising a computer-generated random number sequence. To keep both intervention groups balanced, randomization will be stratified for sex (male versus female) baseline inflammation status (hsCRP<3mg/L versus hsCRP ≥3mg/L) and baseline central sensitization status (central sensitization inventory (CSI) score <40 versus CSI score ≥ 40).
  A list with patient numbers and the group allocation that results from this randomization procedure will be securely stored and only an independent researcher will have direct access to the randomization list. Patients will be scheduled to receive their first assessment within 1 week of randomisation.
  Patients will be recruited in primary care and participating hospitals. Announcements will be placed in newspapers, pharmacies etc.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Outcome assessors will be blinded to the maximal extent possible. With regard to this, patients will be asked not to communicate with the assessors about the intervention received. The researcher who is responsible for the acute measurements, is not blinded for group allocation but the researcher responsible for the basal measurements is. Both researchers are blinded for the outcome analyses. Furthermore, at the end of each assessment, the success of assessor blinding will be examined by asking whether the assessor thought the participant had received the experimental or control intervention, including the percentage of certainty. The physiotherapists providing BGA will not be involved in providing MST, and vice versa. Additionally, the physiotherapists will be blinded for outcome measures. The statistician will be blinded to the allocation of the treatment groups and statistical analyses will be performed in a blinded manner.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Muscle Strengthening Training (MST)-group (Experimental): Subjects allocated to the MST group (n=30) will perform a muscle strengthening training program of 12 weeks.
  Interventions: Other: Muscle Strengthening Training
- Behavioral Graded Activity (BGA)-group (Experimental): Subjects allocated to the BGA group (n=30) will perform a rehabilitation program according to the principles of behavioural graded activity for a period of 12 weeks.
  Interventions: Behavioral: Behavioral graded activity
- Control group (No Intervention): Subjects allocated to the control group (n=30) have to maintain their current life-style and treatment (if any) and to refrain from other new interventions during 24 weeks.

INTERVENTIONS:
Other: Muscle Strengthening Training — Muscle strengthening training will take place for a period of 12 weeks, in which participants will have 36 exercise sessions (18 at the hospital under supervision of a physiotherapist; 18 unsupervised at home) planned. Muscles of the leg (i.e. quadriceps, hip ab- and adductors) will be trained at 3 set of 10 repetitions at 80% of 1RM with the use of elastic bands. 1RM will be assessed at baseline and the exercise intensity will be progressively increased by 10% of 1RM every two sessions from 50 up to 70-80 % of 1RM. Every 6 sessions, the 1RM will be reassessed and the training resistances will be adapted.
  Arms: Muscle Strengthening Training (MST)-group
Behavioral: Behavioral graded activity — Subjects will receive a behavioural treatment integrated within the concepts of operant conditioning with exercise therapy for a period of 12 weeks, in which the subjects will have maximum 36 BGA sessions (min. 13- max. 18 at the hospital under supervision of a physiotherapist; 18 unsupervised at home) planned. The purpose of BGA is to increase the level of activities in a time-contingent manner and increase the level of physical activity in the subject's daily lives. BGA consists of 3 phases: pain education (phase 1), treatment phase in which subjects increase their level of activity gradually (phase 2) and integration of learned principles in daily live (phase 3).
  Arms: Behavioral Graded Activity (BGA)-group

SUMMARY:
International guidelines recommend exercise as the first choice treatment for knee osteoarthritis (KOA). Muscle strengthening training (MST) and behavioural graded activity (BGA) show comparable effects on KOA pain, but the mechanisms of action are unclear. Understanding these mechanisms is necessary to tailor exercise therapy towards specific mediators and thereby optimize treatment effects. Based on previous studies, both exercise-induced anti-inflammation and endogenous analgesia are promising pathways for pain reduction after exercise therapy. This study aims to examine (anti)-inflammation and endogenous analgesia as mediators for the effect of MST and/or BGA on pain in patients with KOA. Therefore, a 3-arm randomized clinical trial is established: 12 weeks of muscle strengthening training, behavioural graded activity or control. Mediator analysis will be performed. Unravelling the mechanisms of action of exercise therapy in KOA will not only be extremely valuable for researchers, but also for exercise immunology and pain scientists. The results of this research will also find their way into clinical practice: thanks to the current project, tailoring exercise therapy programs towards specific mechanistic factors and thereby optimizing treatment effects will be at the horizon for patients suffering from KOA.

ELIGIBILITY:
Inclusion Criteria:

1. KOA according to the clinical American College of Rheumatology (ACR) criteria. The clinical ACR criteria for KOA are: knee pain and at least 3 of the 6 following features: age ≥50, morning stiffness <30 minutes, crepitus, bony tenderness, bony enlargement, no palpable warmth. KOA will be confirmed with radiographs, including anterior-posterior (AP) and medio-lateral (ML) radiographs for imaging the tibiofemoral joint, and an axial view for imaging the patellofemoral joint. Kellgren and Lawrence (K&L) grading system for OA will be applied, with K&L grade 2 or higher defined as OA; radiographic KOA is defined as definite osteophytes and possible joint space narrowing.
2. pain, nominated by the patient as 3 /10 or higher on a visual analogue scale on most days of the last 3 months
3. aged ≥ 50 years.

Exclusion Criteria:

1. treatment with exercise therapy or joint infiltrations (e.g., corticosteroids, hyaluronic acid) in the preceding 6 months;
2. being on a waiting list for knee replacement;
3. any contra-indication for exercise therapy as established by the treating physician;
4. corticosteroid infiltrations in the last 6 months;
5. cognitive impairment (unable to understand the test instructions and/or Mini Mental State Examination score <23/30);
6. unable to understand the Dutch language;
7. inflammation unrelated to OA (e.g. due to acute or chronic infection) established by CRP>10mg/L.
8. presence of a disorder and/or medication that influences pain and/or the immune system

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Knee pain as primary study outcome | Baseline
  Pain is the primary outcome as it is the primary and most disabling symptom in OA. The pain subscale of the WOMAC Osteoarthritis Index LK3.0 questionnaire will be used for the assessment of pain severity. The Knee injury and Osteoarthritis Outcome Score (KOOS) includes WOMAC Osteoarthritis Index LK3.0 in its complete and original format (with permission). WOMAC (and therefore the pain and symptoms subscale of the KOOS) is a valid tool for subjects with KOA. The KOOS is proven to generate valid and reliable scores.
Knee pain as primary study outcome | during intervention: week 2 (acute)
  Pain is the primary outcome as it is the primary and most disabling symptom in OA. The pain subscale of the WOMAC Osteoarthritis Index LK3.0 questionnaire will be used for the assessment of pain severity. The Knee injury and Osteoarthritis Outcome Score (KOOS) includes WOMAC Osteoarthritis Index LK3.0 in its complete and original format (with permission). WOMAC (and therefore the pain and symptoms subscale of the KOOS) is a valid tool for subjects with KOA. The KOOS is proven to generate valid and reliable scores.
Knee pain as primary study outcome | during intervention: week 10 (acute)
  Pain is the primary outcome as it is the primary and most disabling symptom in OA. The pain subscale of the WOMAC Osteoarthritis Index LK3.0 questionnaire will be used for the assessment of pain severity. The Knee injury and Osteoarthritis Outcome Score (KOOS) includes WOMAC Osteoarthritis Index LK3.0 in its complete and original format (with permission). WOMAC (and therefore the pain and symptoms subscale of the KOOS) is a valid tool for subjects with KOA. The KOOS is proven to generate valid and reliable scores.
Knee pain as primary study outcome | post-intervention: week 13
  Pain is the primary outcome as it is the primary and most disabling symptom in OA. The pain subscale of the WOMAC Osteoarthritis Index LK3.0 questionnaire will be used for the assessment of pain severity. The Knee injury and Osteoarthritis Outcome Score (KOOS) includes WOMAC Osteoarthritis Index LK3.0 in its complete and original format (with permission). WOMAC (and therefore the pain and symptoms subscale of the KOOS) is a valid tool for subjects with KOA. The KOOS is proven to generate valid and reliable scores.
Knee pain as primary study outcome | post-intervention: week 26
  Pain is the primary outcome as it is the primary and most disabling symptom in OA. The pain subscale of the WOMAC Osteoarthritis Index LK3.0 questionnaire will be used for the assessment of pain severity. The Knee injury and Osteoarthritis Outcome Score (KOOS) includes WOMAC Osteoarthritis Index LK3.0 in its complete and original format (with permission). WOMAC (and therefore the pain and symptoms subscale of the KOOS) is a valid tool for subjects with KOA. The KOOS is proven to generate valid and reliable scores.
Knee pain as primary study outcome | post-intervention: week 64
  Pain is the primary outcome as it is the primary and most disabling symptom in OA. The pain subscale of the WOMAC Osteoarthritis Index LK3.0 questionnaire will be used for the assessment of pain severity. The Knee injury and Osteoarthritis Outcome Score (KOOS) includes WOMAC Osteoarthritis Index LK3.0 in its complete and original format (with permission). WOMAC (and therefore the pain and symptoms subscale of the KOOS) is a valid tool for subjects with KOA. The KOOS is proven to generate valid and reliable scores.

SECONDARY OUTCOMES:
Different subtypes of pain: pain | Baseline, during intervention (week 2 and 10), post-intervention (week 13, 26 and 64)
  Pain will be measured using the Visual analogue scale (VAS).
Different subtypes of pain: intermittent pain | Baseline, during intervention (week 2 and 10), post-intervention (week 13, 26 and 64)
  Intermittent pain will be measured using a short and easily applicable self-reported measure, i.e. intermittent and constant pain (ICOAP).
Different subtypes of pain: constant pain | Baseline, during intervention (week 2 and 10), post-intervention (week 13, 26 and 64)
  Constant pain, will be measured using a short and easily applicable self-reported measure, i.e. Intermittent and constant pain (ICOAP).
Different subtypes of pain: central sensitization | Baseline, during intervention (week 2 and 10), post-intervention (week 13, 26 and 64)
  Central sensitization will be measured using an easily applicable self-reported measure i.e. Central Sensitization Inventory (CSI).
Function in daily living (KOOS subscale) | Baseline, post-intervention (week 13, 26 and 64)
  Function in daily living will be measured using self-reported measures. The KOOS function in daily living (ADL) subscale and functioning in sports and recreation subscale are reliable and valid scales to measure function in people with osteoarthritis. The patient global assessment (PGA) is a recommended questionnaire in clinical trials of rehabilitation interventions for OA and it measures the improvement or deterioration of their condition.
Function in daily living (PGA) | Assessed at baseline and post-intervention (at week 13, 26 and 64)
  Function in daily living will be measured using self-reported measures. The patient global assessment (PGA) is a recommended questionnaire in clinical trials of rehabilitation interventions for OA and it measures the improvement or deterioration of their condition.
Treatment adherence | During the intervention (week 1-12) and at week 13
  Patient adherence for the treatment sessions will be calculated as the ratio of the number of treatment sessions that were actually carried out versus the number of prescribed sessions. Compliance will be calculated as the ratio of the total training duration (recorded in the logbooks) versus the prescribed total training duration, multiplied by 100.
Treatment compliance | During the intervention (week 1-12) and at week 13
  Compliance will be calculated as the ratio of the total training duration (recorded in the logbooks) versus the prescribed total training duration, multiplied by 100.
Health care cost effectiveness | Assessed at baseline, at week 13, 26 and 64
  Medical consumption, the type, dose, method of administration and frequency of analgesic, NSAID or symptom-modifying medication, as well as surgeries (total or partial knee replacements) will be recorded. Health care use will be evaluated using the combination of three questionnaires: (1) the Medical Consumption Questionnaire (2) the Productivity Cost Questionnaire and (3) the EuroQol EQ-5D.

OTHER OUTCOMES:
Pain catastrophizing (explanatory outcome) | Assessed at baseline, at week 13, 26 and 64
  Pain catastrophizing will be assessed using the Pain Catastrophizing Scale (PCS-DV).
Pain hypervigilance (explanatory outcome) | Assessed at baseline, at week 13, 26 and 64
  Pain hypervigilance will be assessed using the Pain Vigilance and Awareness Questionnaire (PVAQ).
Illness perceptions (explanatory outcome) | Assessed at baseline, at week 13, 26 and 64
  Illness perceptions will be assessed using the Illness Perception Questionnaire-revised (IPQ-R).
Dietary intake (explanatory outcome) | Assessed at baseline, at week 13, 26 and 64
  Dietary intake will be assessed with the use of the Food Frequency Questionnaire (FFQ).
Inflammation (as treatment mediator) | Assessments will be performed at baseline, during intervention (at week 2 or week 3 and at week 10 or week 11; pre- and post-treatment for the acute effects), at week 13 (at least 48 hours after the last intervention) and at week 64
  Inflammation will be tested by a blood-based biomarker panel (e.g. ELISA) for chronic low-grade inflammatory profile.
Endogenous analgesia as treatment mediator: electrical detection threshold | Assessments will be performed at baseline, during intervention (at week 2 or week 3 and at week 10 or week 11; pre- and post-treatment for the acute effects), and at week 13 (at least 48 hours after the last intervention) and week 64
  Endogenous pain modulation will be evaluated by determining the electrical detection threshold. Electrical stimulation (Surpass LT Stimulator) will start at 0mA and will be gradually increased until the patient is experiencing a faint sensation.
Endogenous analgesia as treatment mediator: electrical pain threshold | Assessments will be performed at baseline, during intervention (at week 2 or week 3 and at week 10 or week 11; pre- and post-treatment for the acute effects), and at week 13 (at least 48 hours after the last intervention) and at week 64
  Endogenous pain modulation will be evaluated by determining the electrical pain threshold. Electrical stimulation (Surpass LT Stimulator) will start at 0 mA and will be gradually increased until the patient is experiencing the stimulus as painful.
Endogenous analgesia as treatment mediator: temporal summation | Assessments will be performed at baseline, during intervention (at week 2 or week 3 and at week 10 or week 11; pre- and post-treatment for the acute effects), at week 13 (at least 48 hours after the last intervention) and at week 64
  Endogenous pain facilitation will be evaluated by the temporal summation paradigm. Electrical stimuli (Surpass LT Stimulator) will be given at the intensity (mA) of the electrical pain threshold. A verbal numeric rating scale (VNRS) from 0 to 10 will be asked at the first stimulus, at the middle and at the last electrical stimulus.
Endogenous analgesia as treatment mediator: conditioned pain modulation | Assessments will be performed at baseline, and at week 13 (at least 48 hours after the last intervention) and at week 64.
  The efficacy of endogenous analgesia will be evaluated by the conditioned pain modulation paradigm. Conditioned pain modulation will be tested with the electrical stimulator as test stimulus and the cold pressor (12 °C) as conditioning stimulus. The difference between the electrical pain threshold (baseline) and the electrical pain threshold during the cold pressor (baseline + cold pressor) is called the conditioned pain modulation effect. After electrical stimulation (Surpass LT Stimulator), a VNRS score from 0 to 10 will be asked.
Endogenous analgesia as treatment mediator: offset-analgesia | Assessments will be performed at baseline and at week 13 (at least 48 hours after the last intervention) and at week 64.
  Endogenous analgesia will be assessed by offset analgesia. Offset analgesia can be described as the disproportionately large decrease in perceived pain following slight decreases in electrical intensity.
  Painful electrical stimuli (Surpass LT Stimulator) will be given to the patients into 3 time intervals. The electrical intensity of time interval 1 and 3 will be the same, while the electrical intensity of time interval 2 will be higher. Participants need to report their intensity of pain according to the visual analogue scale ranging from 0 to 10 during the 3 intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Bautmans, PhD, Principal Investigator — Gerontology department (GERO) and Frailty in Ageing (FRIA) research department, Vrije Universiteit Brussel (VUB), Laarbeeklaan 103, B-1090 Brussels, Belgium
Locations (1):
- Vrije Universiteit Brussel (VUB), Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beckwee D, Nijs J, Bierma-Zeinstra SMA, Leemans L, Leysen L, Puts S, Rice D, Schiphof D, Bautmans I. Exercise therapy for knee osteoarthritis pain: how does it work? A study protocol for a randomised controlled trial. BMJ Open. 2024 Jan 10;14(1):e074258. doi: 10.1136/bmjopen-2023-074258. PMID 38199628